CLINICAL TRIAL: NCT01545505
Title: Early Diagnosis of Risk of Post-Traumatic Stress Disorder (PTSD) Relapse in Children and Their Families
Brief Title: Identification of Markers of Post-Traumatic Stress Disorder (PTSD) Relapse
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 11-AOI-09
Record Dates: First submitted 2011-12-08; First posted 2012-03-06 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Post Traumatic Stress Disorder (PTSD)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- In remission phase of PTSD (Other): Patients having suffered from PTSD in the past and in remission od PTSD and their parents
  Interventions: Behavioral: Neuropsychological assessment
- Activ PTSD (Other): patients suffering from PTSD (Post-traumatic Stress Disorder) and their parents
  Interventions: Behavioral: Neuropsychological assessment

INTERVENTIONS:
Behavioral: Neuropsychological assessment — A clinical evaluation with Impact of Events Scale-Revised, Child Post-Traumatic Stress Reaction Index, State-Trait Anxiety Inventory for Children, Children Depression Inventory and Emotion, activity and sociability.
  A neuropsychological assessment with a emotional Go-No/Go, a visual search task, the Trail Making Test, 3 items of the WISC III ( and the Grober and Buschke Test.

SUMMARY:
Relapse of post-traumatic stress disorder (PTSD) remains challenging. In addition, factors predicting PTSD relapse are still unknown. The aim of this study is to examine whether clinical and neuropsychological changes (e.g., attentional bias toward aversive cues) that characterized PTSD can be observed in people with past PTSD (children and their families) and whether these persistent changes are predictive of PTSD relapse.

DETAILED DESCRIPTION:
One of the great challenges in Psychotraumatology is the high risk (20-40%) of post-traumatic stress disorder (PTSD) relapse, which markers remain understudied. Identification of these markers is of particular interest for the development of strategies to prevent relapse. Based on clinical and experimental data, it appears that (i) the so-called residual clinical symptoms (such as sleep disturbance, irritability) and (ii) the neuropsychological dysfunctions (cognitive difficulties), persisting after remission, may constitute markers of PTSD relapse. Moreover, all of these potential markers have also been linked with dysfunctions, persisting or reoccurring, in the prefrontal cortex after remission.

The main objective of this study is to identify these clinical and neuropsychological markers of PTSD relapse in children and their families. The secondary objective is to demonstrate the link between prefrontal dysfunctions and relapse.

This longitudinal study will include 4 experimental groups:

* 30 children with PTSD
* 30 children with past PTSD (children in remission)
* 30 parents of children with PTSD
* 30 parents of children with past PTSD The first visit is planned during the symptomatic phase (T0). The second visit (T1) is planned at the end of the symptomatic phase (or 6 months later T0). The last visit is planned 3-months after T1.

The psychological assessment will include:

A structured interview with a psychiatrist An assessment of PTSD symptoms (IES-R, CPTS-RI for children) An assessment of the co-morbidity (STAI C and CDI for children, STAI A-B, BDI for adults).

An evaluation of the social life (EAS for children and SAS-SR for adults).

The neuropsychological assessment will include:

An evaluation of the attentional treatment (Go-No / go and visual search) An evaluation of executive functions (TMT A and B) A brief evaluation of the IQ (items memory of figures, matrix and resemblance) An evaluation of the memory (Grober and Buschke) Tests include an adult and children versions that are validated. All studies will be conducted at the Nice University Hospital, Tours University Hospital and Toulouse University Hospital.

ELIGIBILITY:
For children

Inclusion Criteria:

* Children (9/18 years)
* Patients who have lived a traumatic event (physical assault and road accident) and who have a PTSD.
* French speaker.
* Participants must sign the informed consent and they must be affiliated to the social insurance.

Exclusion Criteria

* Children who have a neurological pathology.
* Children who have brain damage or brain-injured
* Subject having participated in a biomedical research in three months preceding the inclusion

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-10 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Attentional score | baseline at the first visit (T0), at 6 months, at 9 months
  Go-No/Go and visual search tests

SECONDARY OUTCOMES:
memory (Grober and Buschke) | baseline at the first visit (T0), at 6 months, at 9 months
  Grober and Buschke memory tests

CONTACTS AND LOCATIONS:
Overall Officials: Michel BENOIT, M.D.,PhD, Principal Investigator — Psychiatrie, Hôpital Pasteur, CHU de NICE; Wissam EL HAGE, M.D, PhD, Principal Investigator — Psychiatrie, CHU de TOURS; Frédérique JOVER, M.D., Principal Investigator — CAP, Hôpital St ROCH, CHU de NICE; Florence ASKENAZY, M.D., Principal Investigator — Fondation Lenval, NICE; Philippe BIRMES, M.D., Principal Investigator — Psychiatrie, CHU de TOULOUSE; Virginie BUISSE, M.D., Principal Investigator — CAP, Hôpital St Roch, CHU de NICE
Locations (4):
- France (4):
  - CHU de NICE, Nice
  - Fondation Lenval, Nice
  - CHU de TOULOUSE, Toulouse
  - CHU de TOURS, Tours